CLINICAL TRIAL: NCT00914186
Title: A Multicenter, Randomized, Double-Blind, Vehicle-Controlled Study of the Efficacy, Safety and Tolerability of TS-022 in Adult Patients With a Diagnosis of Atopic Dermatitis (AD) With Moderate to Very Severe Pruritus
Brief Title: Study of TS-022 in Adult Patients With Atopic Dermatitis With Pruritus (POC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taisho Pharmaceutical R&D Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TS022-US201
Record Dates: First submitted 2009-05-28; First posted 2009-06-04 (Estimated); Results first posted 2011-11-17 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Pruritus
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle
- TS-022 0.005% lotion (Experimental)
  Interventions: Drug: TS022
- TS-022 0.010% lotion (Experimental)
  Interventions: Drug: TS022
- TS-022 0.020% lotion (Experimental)
  Interventions: Drug: TS022

INTERVENTIONS:
Drug: TS022 — Lotion
  Arms: TS-022 0.005% lotion; TS-022 0.010% lotion; TS-022 0.020% lotion
Drug: Vehicle — Lotion
  Arms: Vehicle

SUMMARY:
The purpose and (primary) objectives of this study are to evaluate the efficacy, safety, and tolerability of TS-022 in adults with atopic dermatitis who have moderate to very severe pruritus (itching), following a 28-day regimen of twice-daily topical application.

DETAILED DESCRIPTION:
(none provided)

ELIGIBILITY:
Inclusion Criteria:

1. Adults, males or females, 18 - 65 years of age at the time of obtaining the written Informed Consent
2. Generally healthy subjects, who have no past or present history of any significant and/or newly-diagnosed disease or condition
3. A score of 2 (Mild Disease), 3 (Moderate Disease) or 4 (Severe Disease) on the Investigator's Global Assessment of Atopic Dermatitis (IGA) Scale
4. A score of 2 (Moderate Pruritus), 3 (Severe Pruritus) or 4 (Very Severe Pruritus) on the Five-Point Pruritus Scale
5. Patient satisfies the diagnostic criteria for AD as determined by the criteria of Hanifin and Rajka
6. Patient understands the study procedures and agrees to participate in the study by giving written Informed Consent
7. Ability to read and understand English and to provide written informed consent and authorization for protected health information disclosure

Exclusion Criteria:

1. Concurrent skin pathology or recent history (within the past 5 years) of a chronic skin disease other than AD
2. Use of phototherapy, including exposure to tanning beds, within 28 days of Study Drug application
3. Taking systemic immunosuppressive drugs, biologicals, or corticosteroids therapy within (14 days), or topical immunosuppressive drugs or corticosteroid therapy (within 7 days) of Study Drug application
4. Females who are planning a pregnancy, who are pregnant, or who are breastfeeding
5. Inability or unwillingness to discontinue current AD treatment(s)
6. Inability or unwillingness to comply with study visit schedule and/or other study activities as required by the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nermina Nakas, MD, Study Director — Clinsys
Locations (15):
- United States (15):
  - UCSD, La Jolla, California
  - Therapeutics Clinical Research, San Diego, California
  - Ameriderm Research, Jacksonville, Florida
  - Ameriderm Research, Kissimmee, Florida
  - FXM Research, Miramar, Florida
  - Ameriderm Research, Ormond Beach, Florida
  - Gwinnett Clinical Research, Snellville, Georgia
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Wake Forest University, Winston-Salem, North Carolina
  - Haber Dermatology and Cosmetic Surgery, Inc, South Euclid, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - J & S Studies, College Station, Texas
  - Center for Clinical Studies, Houston, Texas
  - Center for Clinical Studies, Webster, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period for the study started 03Jun09. It was the responsibility of the PI for advertisement and recruitment of the study.
Pre-assignment Details: There was a seven day run-in-period in which subjects self-applied the Vehicle control twice daily.
Groups:
- Vehicle: once daily
- TS-022 0.005%; TS-022 0.010%; TS-022 0.020%: lotion/once daily
Period: Overall Study
Arm/Group | Vehicle | TS-022 0.005% | TS-022 0.010% | TS-022 0.020%
Started | 31 | 30 | 31 | 30
Completed | 28 | 28 | 29 | 20
Not Completed | 3 | 2 | 2 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle | TS-022 0.005% | TS-022 0.010% | TS-022 0.020% | Total
Number analyzed (Participants) | 31 | 30 | 31 | 30 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 30 | 31 | 30 | 122
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.5 (13.53) | 38.0 (11.63) | 35.1 (13.78) | 39.0 (13.89) | 36.4 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 17 | 20 | 77
  Male | 12 | 9 | 14 | 10 | 45
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 31 | 30 | 122

OUTCOME MEASURES:

1. Primary Outcome: Change in Pruritis Visual Analog Scale (VAS)
Description: Patient reported outcome of pruritis measurement (0-100 mm/min-max)on a change in visual analog scale
Time Frame: Baseline through Study Day 36 (Visit 7)
Population: Intent To Treat (ITT) analysis
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Vehicle | TS-022 0.005% | TS-022 0.010% | TS-022 0.020%
Number analyzed (Participants) | 29 | 28 | 29 | 21
mm | -12.4 (14.09) | -15.5 (18.38) | -13.9 (21.11) | -6.2 (18.82)

2. Primary Outcome: Safety and Tolerability of TS-022 Topical Lotion as Measured by Participants Who Demonstrated Adverse Events
Description: Safety assessment of all subjects who received investigational product. Outcome measure is number of subjects with an adverse event. Measures of adverse events in participants included vital signs, laboratory findings, physical exams, electrocardiograms
Time Frame: Baseline through Study Day 36 (Visit 7)
Population: total number of subjects who received study drug.
Measure: Number; unit: participants
Arm/Group | Vehicle | TS-022 0.005% | TS-022 0.010% | TS-022 0.020%
Number analyzed (Participants) | 31 | 30 | 30 | 31
participants | 9 | 11 | 10 | 11

3. Primary Outcome: Investigator's Global Assessment (IGA) Based on a Dermatologist's Evalution of the Change in Subject's Score of Target Treatment Areas
Description: investigator assessment of disease status rated on 0-5 scale (0 = clear to 5 = very severe) based on a change in score from baseline to Study Day 36 (Visit 7)
Time Frame: baseline through Study Day 36 (Visit 7)
Population: ITT
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Vehicle | TS-022 0.005% | TS-022 0.010% | TS-022 0.020%
Number analyzed (Participants) | 29 | 28 | 29 | 21
units on a scale | -0.6 [-0.9 to -0.3] | -0.5 [-0.8 to -0.2] | -0.6 [-0.8 to -0.2] | -0.6 [-0.8 to -0.2]

4. Primary Outcome: Five Point Pruritus Scale for Self-Assessment of Target Treatment Area Based on a Change in Score
Description: self-assessment using a five point scale of pruritus state based on a change in scale from none (0) to very severe (4), interfering with daily or sleep activities. Subjects will complete the Five-Point Pruritus Scale once at Screening (Visit 1), then twice daily beginning at baseline, which occurs on the morning of Study Day -7 (Visit 2), through Study Day 36 (Visit 7)
Time Frame: Baseline, which is Day -7 (Visit 2), through Day 36 (Visit 7)
Population: ITT
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Vehicle | TS-022 0.005% | TS-022 0.010% | TS-022 0.020%
Number analyzed (Participants) | 29 | 28 | 29 | 21
units on a scale | -0.4 [-0.7 to -0.2] | -0.5 [-0.6 to -0.1] | -0.6 [-0.9 to -0.3] | -0.2 [-0.5 to -0.1]

5. Primary Outcome: Eczema Area and Severity Index (EASI) Based on a Change in Score of Eruption in Proportionate Body Surface Areas
Description: The head and neck [10%], trunk [30%], upper extremities [20%] and lower extremities [40%] were assessed separately for erythema (E), infiltration/papulation (I), excoriation (Ex) and lichenification (L) represented by a numeric coded value of (0, No eruption) to (6, 90% - 100% eruption). One score given to each part of the body on a scale from 1-6 based on the four attributes (E, I, Ex, L) and then a proportional average is taken to get a total score of 1-6.
Time Frame: baseline through Study Day 36 (Visit 7)
Population: ITT analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle | TS-022 0.005% | TS-022 0.010% | TS-022 0.020%
Number analyzed (Participants) | 29 | 28 | 29 | 21
units on a scale | -3.1 (4.75) | -2.1 (5.09) | -2.7 (3.87) | -2.3 (4.50)

6. Primary Outcome: Skindex-29 Questionnaire to Measure the Subject's Overall Quality of Life Based on Activities of Daily Living That Affect Change in Emotion (10 to 50 Points), Symptoms (7 to 35 Points) and Functioning (12 to 60 Points) to Skin Over One Week Period.
Description: Assessment of subject's activities of daily living using the SKINDEX-29 questionnaire to measure the subject's overall quality of life based on a change in scale from baseline. The SKINDEX scoring scale has a range of 29-145. The smaller the number the better the patient feels. The results are the difference of the SKINDEX scoring scale at treatment discharge (day 22) minus baseline (day-7). Hence the results should be negative, as the patient's emotion, symptoms and functioning of the skin should feel better at treatment discharge as opposed to baseline.
Time Frame: Study Day -7 through Study Day 22
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle | TS-022 0.005% | TS-022 0.010% | TS-022 0.020%
Number analyzed (Participants) | 31 | 30 | 30 | 29
units on a scale | -11.7 (11.61) | -12.1 (14.79) | -12.3 (17.56) | -4.1 (12.43)

7. Primary Outcome: Number of Participants Who Had Measurable Pruritis Based on a Visual Horizontal Analog Scale
Description: Pruritis Visual Analog Scale (VAS) based on patient reported outcome of pruritis measurement on a VAS indicating the amount of pruritus (itchiness) experienced from the time of last dose application through the time just before current dose application. Change in pruritus is assessed twice daily beginning at baseline, Study Day -7 (Visit 2), through Study Day 36 (Visit 7). Subjects determine measurable pruritis using a visual horizontal analog scale ranging from "No Itch", even the slightest itch or "Slight Itch", to "Worst Itch Imaginable" to denote the increase in severity of itching.
Time Frame: Baseline through Study Day 36 (Visit 7)
Measure: Number; unit: participants
Groups:
- TS-022: lotion/once daily
Arm/Group | Vehicle | TS-022
Number analyzed (Participants) | 29 | 78
participants | 29 [12.4 to 14.09] | 78 [15.5 to 18.82]

ADVERSE EVENTS:
Time Frame: Safety and tolerability were assessed daily starting at Study Day -7 (Visit 2) through Study Day 52 (End of Study)
Description: Safety variables for evaluation included:
  * adverse events (AEs)
  * clinical laboratory assessments (blood chemistry, hematology, and urinalysis)
  * vital signs
  * physical examinations
  * electrocardiograms
  * pregnancy testing for females of child-bearing potential at specified times throughout the study
Arm/Group | Vehicle | TS-022 0.005% | TS-022 0.010% | TS-022 0.020%
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 9/31 | 11/30 | 10/31 | 11/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=31) | TS-022 0.005% (N=30) | TS-022 0.010% (N=31) | TS-022 0.020% (N=30)
Stomach Discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (3) | 2 (2) | 1 (2)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 2 (2) | 5 (5)
ECG Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Uppper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Slower than expected enrollment and a higher than expected screen failure rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days